### Infant and Child European Cryoablation Project

ClinicalTrials.gov study ID: 18BB37



CONFIDENTIAL

# Parent/Guardian consent form

Date of most recent review: 16<sup>th</sup> November 2020

Version 2 16/11/2020 1

# Infant and Child European Cryoablation Project

ClinicalTrials.gov study ID: 18BB37



#### CONFIDENTIAL

#### PARENT/GUARDIAN CONSENT FORM

| | Please Initial the Boxes | | |
|---|---|---|---|
| 1. | I confirm that I have read and understand the information sheet(s) dated 05/10/2018 version 1 for the above study, have been informed of the nature, significance, implications and risks associated with it and have had the opportunity to ask questions. | | |
| 2. | I understand that my child's participation is voluntary and that I am free to withdraw at any time, without giving any reason, without his/her medical care or legal rights being affected. | | |
| 3. | I understand that sections of any of my child's medical notes may be looked at by responsible physicians or authorised persons from sponsor organisation, regulatory authorities or hosting organisations where it is relevant to my/my child's taking part in research. I give permission for these individuals to have access to his/her records | | |
| 4. | I agree to take part in the above study. | | |
| 5. I agree that I might be contacted in the future for a long-term follow-up Name of Child: | | | |
| Name of Parent/Guardian | | Date | Signature |
| Relationship with Child | | | |
| Name of person taking consent | | | |
| (if different from Investigator) | | | |
| Name of Investigator | | | |
| Name of Interpreter (if applicable) | | | |

1 copy for patient, 1 for researcher, 1 copy to be kept with hospital notes

Version 2 16/11/2020 2